CLINICAL TRIAL: NCT05413356
Title: Ruxolitinib for Newly Diagnosed Bronchiolitis Obliterans Syndrome After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Ruxolitinib for Newly Diagnosed Bronchiolitis Obliterans Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Sir Run Run Shaw Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other); The Affiliated People's Hospital of Ningbo University (Other Government); Jinhua Central Hospital (Other); Taizhou Hospital (Other); Union hospital of Fujian Medical University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJU-HSCT-BOS
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-05

CONDITIONS: Bronchiolitis Obliterans Syndrome; Hematologic Malignancy
Keywords: Allogeneic Hematopoietic stem cell transplantation; chronic graft versus host disease; bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): Ruxolitinib twice daily treatment, combined with steroids 1mg/kg/day for two weeks, and tampering 0.25 mg/kg/day every week
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Oral ruxolitinib twice daily
  Other Names: Ruxolitinib twice daily

SUMMARY:
Lung is one of the target organs in chronic graft versus host disease (cGVHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT). Bronchiolitis obliterans syndrome (BOS) after allo-HSCT was a clinical syndrome characterized by persistent airflow restriction which is the result of lung cGVHD. BOS is one of the main causes of late mortality after allo-HSCT, severely restricting the daily activities and respiratory function of patients. It limits the quality of life and increased the non-relapse mortality (NRM) after allo-HSCT. Currently, the first-line treatment for BOS is FAM ( oral fluticasone, azithromycin and montelukast). However, more than 50% of patients develop as steroids resistant (SR)-BOS, and SR-BOS has a poor prognosis and irreversible impaired lung function. Ruxolitinib is an effective drug in the treatment of SR-cGVHD. This is a phase Ⅱ prospective clinical study to explore the efficacy and safety of ruxolitinib as a first-line treatment for newly diagnosed BOS after allo-HSCT.

DETAILED DESCRIPTION:
The incidence of chronic graft versus host disease (cGVHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT) was 30%-70%, Which extremely limited the quality of life and the survival of patients after allo-HSCT. Lung is one of the target organs in cGVHD after allo-HSCT. Bronchiolitis obliterans syndrome (BOS) after allo-HSCT was a clinical syndrome characterized by persistent airflow restriction which is the result of lung cGVHD. BOS is one of the main causes of late mortality after allo-HSCT, severely restricting the daily activities and respiratory function of patients. It limits the quality of life and increased the non-relapse mortality (NRM) after allo-HSCT. Currently, the first-line treatment for BOS is FAM ( oral fluticasone, azithromycin and montelukast). However, more than 50% of patients develop as steroids resistant (SR)-BOS, and SR-BOS has a poor prognosis and irreversible impaired lung function. Ruxolitinib is an effective drug in the treatment of SR-cGVHD. This is a phase Ⅱ prospective clinical study to explore the efficacy and safety of ruxolitinib as a first-line treatment for newly diagnosed BOS after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-65 years old
2. Diagnosis of BOS after allo-HCT defined as the 2014 NIH criteria
3. Life expectancy > 6 months at the time of enrollment
4. At least 4 weeks since initiation of the most recent systemic therapy for cGVHD or BOS
5. The ability to understand and willingness to sign a written consent document

Exclusion Criteria:

1. Recurrent malignancy or disease progression requiring anticancer therapy
2. Currently receiving or have previously received ruxolitinib for chronic GVHD therapy
3. Known history of allergy to ruxolitinib or its excipients
4. Hepatic dysfunction: transaminases (ALT, AST) > 5X ULN and/or total bilirubin > 3X ULN
5. Hematologic dysfunction: absolute neutrophil count <1000/μL, platelet cout <30*10E9/L, and/or Hgb < 8 g/dL
6. Renal dysfunction: calculated creatinine clearance < 30 mL/min (Cockcroft-Gault formula)
7. previously received second-line treatment or any drugs in clinical trials for cGVHD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
absolute FEV1 increase | 3 Months
  The proportion of participants with a sustained, absolute FEV1 increase by ≥ 10% after 3 months of treatment with ruxolitinib (compared to baseline measure prior to study enrollment)

SECONDARY OUTCOMES:
treatment failure rate | 3 Months
  The proportion of participants who do not experience a sustained, absolute decrease in FEV1 by ≥ 10% after 3 months of treatment with ruxolitinib (compared to baseline measure prior to study enrollment)
absolute FEV1 increase | 6 Months, 9 Months, 12 Months and 24 Months
  The proportion of participants with a sustained, absolute FEV1 increase by ≥ 10% after treatment with ruxolitinib (compared to baseline measure prior to study enrollment)
Improvements in chronic GVHD organ specific manifestations | 6 Months, 9 Months, 12 Months and 24 Months
  mprovements in chronic GVHD organ specific manifestations will be categorized according to the NIH chronic GVHD consensus criteria.
Overall Survival | 2 years
  The proportion of patients survival at two years after enrollment of ruxolitinib treatment
cGVHD progression-free survival | 2 years
  Participants alive without cGVHD progression are censored at the date of last disease evaluation
The incidence and types of serious adverse events | From the start of treatment until 30 days after the end of treatment, up to 2 years
  Adverse events are graded according to Common Terminology Criteria for Adverse Events (CTCAE v4)
The change of systemic corticosteroid dose over time | From the start of treatment until the end of treatment, up to 2 years
  The change of systemic corticosteroid dose over time during the treatment of BOS

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, M.D., Principal Investigator — First Affilaated Hospital of Medical School of Zhejiang University
Locations (1):
- The first Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No